CLINICAL TRIAL: NCT01402973
Title: Pilot Study of a Dietary Intervention Based Upon Advanced Glycation End Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Collaborators: Johns Hopkins University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Richard Semba, The Johns Hopkins University School of Medicine
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AGE Dietary Intervention
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-AGE Diet (Experimental): The high-AGE diet will be approximately four times higher in AGEs than the low-AGE diet.
  Interventions: Other: Dietary
- Low-AGE Diet (Experimental): The low-AGE diet will be approximately four times lower in AGEs than the high-AGE diet.
  Interventions: Other: Dietary

INTERVENTIONS:
Other: Dietary — The diets will each consist of 3 meals/day and 1 snack/day which are either high or low in AGEs.

SUMMARY:
The purpose of this pilot study is to determine whether it is feasible to conduct a randomized, controlled dietary intervention trial of high versus low dietary intake of advanced glycation end products (AGEs) in 24 adults; and to gather preliminary data on the impact of high versus low AGE diet health parameters. The investigators hypothesize that it will be feasible to conduct a randomized, parallel arm, controlled dietary intervention in a pilot study involving 24 subjects.

DETAILED DESCRIPTION:
Advanced glycation end products (AGEs), bioactive molecules formed by the non-enzymatic glycation of proteins, are emerging as a possible dietary risk factor for many key adverse health outcomes related to obesity and to aging. Major sources of systemic AGEs are endogenous AGEs generated in the body and exogenous AGEs found in foods. When food is heated to high temperatures, the characteristic "browning" generates Maillard reaction products, known as AGEs. Although AGEs have been implicated in atherosclerosis, insulin resistance, diabetes, cardiovascular disease, aging-related eye disease, Alzheimer's disease, and chronic kidney disease, the possible adverse effects of dietary AGEs have not been well characterized in humans.

The objective of the study is to determine whether it is feasible to conduct a randomized, parallel arm, controlled dietary intervention in a pilot study involving 24 subjects; and to compare the effects of a high-AGE and low-AGE diet on (a) serum and urine carboxymethyl-lysine and serum receptor for AGEs (RAGE), (b) endothelial function, (c) interleukin-6, C-reactive protein, (d) lipids, (e) adipokines, (f) glucose metabolism and insulin resistance, (g) renal function, and (h) cognition.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older and less than 70 years of age
* Non-smoker
* Body mass index of 18.5 to <30 mg/kg2

Exclusion Criteria:

* Diabetes, thyroid disease, angina, myocardial infarction, heart failure, stroke, peripheral artery disease, chronic obstructive pulmonary disease, inflammatory bowel disease, liver disease, chronic kidney disease, or Raynaud's disease
* Taking regular vitamin supplements, or if taking regular vitamin supplements, not willing to discontinue taking vitamin supplements while participating in the study
* Taking vitamin B6 (pyridoxamine) supplements (50 mg or more)
* Taking aspirin or nonsteroidal anti-inflammatory medications (NSAIDS), or if so, not willing to discontinue taking aspirin or NSAIDS while participating in the study
* Major food allergies (i.e., dairy, nuts, etc)
* History of eating disorders or other dietary patterns that are not consistent with the dietary intervention (e.g. vegetarians, very low fat diets, high protein diets)
* Loss of 10% of body weight within the last 12 months or plan to initiate a weight loss program during the next two months
* Self-report of alcohol or substance abuse with the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the study doctor may interfere with study participation or the ability to follow the intervention protocol
* Not willing to consume the diets being tested by the study
* Cognitive impairment, indicated by a Mini-Mental State Exam score <23
* Triglycerides >300 mg/dL
* Hemoglobin ≤11 g/dL
* Creatinine greater or equal to 1.5 mg/dL
* Fasting plasma glucose >125 mg/dL
* Proteinuria
* Long fingernails on the index finger of each hand, or if so, not willing to trim these two fingernails so that peripheral arterial tonometry can be conducted during the study
* Not willing to give written, informed consent to participate in the study
* Women who are lactating or pregnant, or plan to become pregnant during the study

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Endothelial function | At baseline and following 6-week intervention
  Endothelial function will be measured using peripheral arterial tonometry.
Biomarkers | At baseline and following 6-week intervention
  Fasting venous blood samples will be drawn for measurements of CML, IL-6, CRP, leptin, adiponectin, cystatin C, cholesterol, triglycerides, glucose, insulin, sRAGE, and esRAGE. Urinary creatinine and CML also will be measured.

SECONDARY OUTCOMES:
Cognitive function and mood | At baseline and following 6-week intervention
  Five cognitive tests and a test of mood will be used to assess various cognitive parameters including attention, memory, and reasoning.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Semba, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Semba RD, Gebauer SK, Baer DJ, Sun K, Turner R, Silber HA, Talegawkar S, Ferrucci L, Novotny JA. Dietary intake of advanced glycation end products did not affect endothelial function and inflammation in healthy adults in a randomized controlled trial. J Nutr. 2014 Jul;144(7):1037-42. doi: 10.3945/jn.113.189480. Epub 2014 Apr 17. PMID 24744309